CLINICAL TRIAL: NCT04980599
Title: Effect of a Probiotic Strain Lactobacillus Paracasei K56 on Metabolic Symptom - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZBao
Record Dates: First submitted 2021-07-08; First posted 2021-07-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Adiposity
Keywords: obesity; lactobacillus paracasei; body fat; visceral fat area
MeSH Terms: conditions — Obesity | interventions — maltodextrin; Probiotics; E 10

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- K56 very high dose -E1 (Active Comparator): Probiotic drink (lactobacillus paracasei K56 10^11CFU) 350ml/d , for 60days
  Interventions: Dietary Supplement: probiotic drink with Lactobacillus paracasei K56
- control -E2 (Placebo Comparator): maltodextrin , for 60days
  Interventions: Dietary Supplement: maltodextrin
- K56 high dose-E3 (Active Comparator): Probiotic powder 1.5g/sachet , 3.0g/d (lactobacillus paracasei K56 10^10cfu) , for 60days
  Interventions: Dietary Supplement: Probiotic powder E3
- K56 middle dose-E5 (Active Comparator): Probiotic powder 8.0g/sachet , 8g/d ( Lactobacillus paracasei K56 10^9cfu) , for 60days
  Interventions: Dietary Supplement: Probiotic powder E5
- K56 low dose -E7 (Active Comparator): probiotic k56 capsule, 2capsules/d ( Lactobacillus paracasei K56 10^7cfu) , for 60days
  Interventions: Dietary Supplement: probiotic capsule E7
- K56 middle dose-E9 (Active Comparator): probiotic K56 capsule, 2capsules/d (Lactobacillus paracasei K56 10^9cfu) ,for 60days
  Interventions: Dietary Supplement: probiotic capsule E9
- K56 high dose-E1K (Active Comparator): probiotic K56 capsule, 2capsules/d (Lactobacillus paracasei K56 10^10cfu), for 60days
  Interventions: Dietary Supplement: probiotic capsule E10
- K56 very high dose-E11 (Active Comparator): probiotic K56 capsule, 4capsules/d (Lactobacillus paracasei K56 10^11cfu) ,for 60days
  Interventions: Dietary Supplement: probiotic capsule E11

INTERVENTIONS:
Dietary Supplement: probiotic drink with Lactobacillus paracasei K56 — Probiotic drink (K56 10^11CFU) 350ml/d for 60days
  Arms: K56 very high dose -E1
Dietary Supplement: maltodextrin — maltodextrin ,for 60days
  Arms: control -E2
Dietary Supplement: Probiotic powder E3 — Probiotic powder 3.0g/d (K56 10^10cfu) 60days;
  Arms: K56 high dose-E3
Dietary Supplement: Probiotic powder E5 — probiotic powder 8g/day for 60days
  Arms: K56 middle dose-E5
Dietary Supplement: probiotic capsule E7 — probiotic k56 capsule, 2capsules/d (10^7cfu) for 60days
  Arms: K56 low dose -E7
Dietary Supplement: probiotic capsule E9 — probiotic k56 capsule, 2capsules/d (10^9cfu) for 60days
  Arms: K56 middle dose-E9
Dietary Supplement: probiotic capsule E10 — probiotic k56 capsule, 2capsules/d (10^10cfu) for 60days
  Arms: K56 high dose-E1K
Dietary Supplement: probiotic capsule E11 — probiotic k56 capsule, 4capsules/d (10^11cfu) for 60days
  Arms: K56 very high dose-E11

SUMMARY:
Recent data suggest that gut microbiota can function as an environmental factor that modulates the amount of body fat and obese individuals have an altered gut microbiota.The results of previous animal studies have suggest that a probiotic strain Lactobacillus paracasei K56 have reduced high-fat diet induced obesity.

In this before-after pilot study, the participants were randomly assigned to 8 groups to compare the fat-reducing effect of the Lactobacillus paracasei K56 by continuously supplementing different product prototypes , and screen the best probiotic K56 prototype with the effect of fat reduction.

ELIGIBILITY:
Inclusion Criteria:

* BMI>=30kg/m2,or percent of body fat(PBF) >=25% for male, >=30 for female.
* Age: 18 - 60 years old adults

Exclusion Criteria:

* patients with severe chronic diseases (coronary heart disease, diabetes, hypertension, immune deficiency, mental disorders, tumors, liver and kidney dysfunction, etc.) and complications;irritable bowel syndrome
* History of intervention with fat-reducing drugs or health products in the past 2 months
* take weight control measures (diet, exercise, etc.) within the past month
* Those who cannot guarantee to maintain their current lifestyle during the trial period
* Those who fail to consume the tested samples as required, or fail to follow up on time, resulting in failure to determine the efficacy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
percent body fat | 60days
  percent body fat (%) will be assessed at baseline and after 60days of intervention
visceral fat area | 60days
  visceral fat area (cm^2) will be assessed at baseline and after 60days of intervention

SECONDARY OUTCOMES:
Serum Lipid Profile | 60 days
  Serum total cholesterol(mmol/L)，Serum triglycerides(mmol/L)，Low-density lipoprotein(mmol/L)，High density lipoprotein(mmol/L) will be measured at baseline and after 60days of intervention
fasting blood glucose | 60 days
  fasting blood glucose(mmol/L) will be measured at baseline and after 60days of intervention
Glycated hemoglobin | 60 days
  Glycated hemoglobin(%) will be measured at baseline and after 60days of intervention
Glycosylated albumin | 60 days
  Glycosylated albumin(%) will be measured at baseline and after 60days of intervention
skeletal muscle mass | 60 days
  skeletal muscle mass (kg) will be assessed at baseline and after 60days of intervention
waist to hip ratio (WHR) | 60 days
  waist to hip ratio (WHR) will be assessed at baseline and after 60days of intervention
Body Mass Index BMI | 60 days
  Body Mass Index (kg/m^2) will be assessed at baseline and after 60days of intervention
body weight | 60 days
  Body weight (kg) will be assessed at baseline and after 60days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ying Feng, Ph.D, Study Director — Hua Dong Hospita Affiliated to Fu Dan University, Shanghai,China
Locations (1):
- Hua Dong Hospital Affiliated to Fu Dan University, Shanghai, China

REFERENCES:
- [Derived] Kadeer G, Fu W, He Y, Feng Y, Liu WH, Hung WL, Feng H, Zhao W. Effect of different doses of Lacticaseibacillus paracasei K56 on body fat and metabolic parameters in adult individuals with obesity: a pilot study. Nutr Metab (Lond). 2023 Mar 21;20(1):16. doi: 10.1186/s12986-023-00739-y. PMID 36944956